CLINICAL TRIAL: NCT04066894
Title: A Phase II Study of Sacral Nerve Stimulation for Low Anterior Resection Syndrome or Fecal Incontinence in Patients Following a Low Anterior Resection or Proctectomy With Coloanal Anastomosis or in Patients After Pelvic Chemoradiation (RESTORE)
Brief Title: Sacral Nerve Stimulation in Treating Low Anterior Resection Syndrome or Fecal Incontinence in Patients With Locally Advanced Rectal Cancer or Other Pelvic Cancer, the RESTORE Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to Issues Enrolling Patients
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-0754; NCI-2019-02649 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0754 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-06-11; First posted 2019-08-26 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Low Anterior Resection Syndrome; Malignant Anal Neoplasm; Malignant Bladder Neoplasm; Malignant Cervical Neoplasm; Malignant Ovarian Neoplasm; Malignant Pelvic Neoplasm; Malignant Prostate Neoplasm; Malignant Uterine Neoplasm; Malignant Vaginal Neoplasm; Malignant Vulvar Neoplasm; Rectal Carcinoma
MeSH Terms: conditions — Low Anterior Resection Syndrome; Anus Neoplasms; Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Ovarian Neoplasms; Pelvic Neoplasms; Prostatic Neoplasms; Uterine Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms; Rectal Neoplasms | interventions — Device Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Supportive Care (sacral nerve stimulator) (Experimental): Patients undergo scheduled, elective surgery for placement of the sacral nerve stimulator with external battery pack. After 2 weeks, patients undergo implantation of a subcutaneous internal battery or removal of the leads if the sacral nerve stimulator is working but does not improve symptoms. If the sacral nerve stimulator is not working, it is repositioned and patients return 2 weeks later for implantation of external battery or removal of leads.
  Interventions: Procedure: Explantation; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Device: Sacral Nerve Stimulator; Device: Sacral Nerve Stimulator Battery; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Procedure: Explantation — Undergo lead removal
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Device: Sacral Nerve Stimulator — Undergo sacral nerve stimulator implantation
  Other Names: Sacral Neuromodulator
Device: Sacral Nerve Stimulator Battery — Undergo sacral nerve stimulator battery implantation
  Other Names: Sacral Neuromodulator Battery
Procedure: Therapeutic Conventional Surgery — Undergo sacral nerve stimulator implantation

SUMMARY:
This phase II trial studies how well sacral nerve stimulation works in treating low anterior resection syndrome or fecal incontinence (the body's passage of stool without control) in patients with rectal cancer that has spread to nearby tissues or lymph nodes, or other pelvic cancer. Sacral nerve stimulation is a permanent implant that may improve bowel functions by stimulating the nerves that control the muscles related to bowel function.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the efficacy of sacral nerve stimulator placement in patients with fecal incontinence (FI) or low anterior resection syndrome (LARS) who have previously undergone chemoradiation treatment (XRT) and/or a restorative partial or complete proctectomy with colorectal or coloanal anastomosis for cancer treatment as per standard of care (restorative surgery cohort).

II. To evaluate the feasibility of sacral nerve stimulator placement in patients with fecal incontinence (FI) or other defecatory dysfunction who have received pelvic radiation treatment without undergoing rectal or other pelvic surgery as per standard of cancer care (radiation only cohort).

SECONDARY OBJECTIVES:

I. To evaluate the effectiveness of sacral nerve stimulation (SNS) as measured by validated questionnaires in patients with FI or LARS within both patient cohorts.

II. To evaluate pelvic floor and sphincter physiology using anorectal manometry (ARM) before and after SNS in patients with FI or LARS within both patient cohorts.

III. To assess potential impact of SNS on urinary incontinence measuring a post-void urinary bladder residual and validated urinary symptom questionnaires in both patient cohorts.

IV. To assess efficacy of SNS on long-term bowel dysfunction at 1 and 3 years post battery implantation as measured by validated questionnaires for both patient cohorts.

OUTLINE:

Patients undergo scheduled, elective surgery for placement of the sacral nerve stimulator with external battery pack. After 2 weeks, patients undergo implantation of a subcutaneous internal battery or removal of the leads if the sacral nerve stimulator is working but does not improve symptoms. If the sacral nerve stimulator is not working, it is repositioned and patients return 2 weeks later for implantation of external battery or removal of leads.

After completion of study, patients are followed up at 1 month, 1 year, and 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: Patients with pathologically proven diagnosis of primary rectal cancer
* Cohort 1: Patients who have previously undergone surgical resection and anastomosis (restorative) with curative intent treatment with or without chemoradiation
* Cohort 1: Patients treated with restorative surgical resection without radiation
* Cohort 1: Patients with any T-stage or N-stage rectal cancer that underwent treatment with radiation and restorative surgery
* Cohort 1: Patients with self-reported FI or LARS
* Cohort 1: Patients must be at least 18 years old and be able to speak and understand English
* Cohort 1: Patients must be willing to and able to sign an approved informed consent document
* Cohort 1: Patients must be >= 24 months post-resection of rectal cancer
* Cohort 1: Patients must have failed prior conservative measures such as Metamucil and motility medications and already been assessed and treated in a pelvic floor rehabilitation program (biofeedback) designed to treat FI and LARS, and continue to experience significant defecatory dysfunction, allowable per principal investigator (PI) discretion
* Cohort 1: Patients must be willing and able to complete Patient Reported Outcomes Questionnaires for before device placement, during the testing phase following lead placement, and after implantation of the battery
* Cohort 1: Patients must be willing and able to undergo elective ARM testing to objectively measure pelvic floor function
* Cohort 1: Patients who have an average resting tone < 40 mmHg (normal > 40 mmHg) and maximal tolerance < 200 milliliters (normal 200-300 milliliters) as measured by ARM
* Cohort 2: Patients with pathologically proven malignancy of the pelvis, other than rectal cancer (e.g. prostate, bladder, anus, vagina, vulva, cervix, uterus, or ovary)
* Cohort 2: Patients treated with standard of care radiation therapies without surgical resection
* Cohort 2: Patients with self-reported FI or other defecatory dysfunction
* Cohort 2: Patients must be at least 18 years old and be able to speak and understand English
* Cohort 2: Patients must be willing to and able to sign an approved informed consent document
* Cohort 2: Patients must be >= 18 months post-pelvic chemoradiation
* Cohort 2: Patients must have already been assessed and treated in a pelvic floor rehabilitation program design to treat FI or other defecatory dysfunction and continue to experience significant defecatory dysfunction
* Cohort 2: Patients must be willing and able to complete Patient Reported Outcomes (PROs) and bowel and bladder diaries (Medtronic) at multiple times during the study
* Cohort 2: Patients must be willing and able to undergo elective ARM testing to measure pelvic floor function
* Cohort 2: Patients who have an average resting tone < 40 mmHg (normal > 40 mmHg) and maximal tolerance < 200 milliliters (normal 200-300 milliliters) as measured by ARM

Exclusion Criteria:

* Cohort 1: Patients with co-morbid illnesses or concurrent disease, which in the judgment of the clinician obtaining informed consent, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Cohort 1: Any diverting bowel ostomy at the time of consent to this study
* Cohort 1: Patients with an absolute neutrophil count (ANC) < 1.7 within 30 days of consent
* Cohort 1: Patients with an international normalized rate (INR) > 1.3 within 30 days of consent
* Cohort 1: Patients with a platelet count < 50 K within 30 days of consent
* Cohort 1: Patients currently being treated with chemotherapy or within preceding 30 days at the time consent
* Cohort 1: Patients previously treated with a SNS for urinary or FI
* Cohort 1: Patients who were documented to have an anastomotic leak following their restorative surgical resection
* Cohort 1: Patients with an Eastern Cooperative Oncology Group (ECOG) performance status > 2 at the time of consent
* Cohort 1: Patients with an active infection requiring systemic therapy at the time of consent
* Cohort 1: Patients with a significant history of uncontrolled cardiac disease including, but not limited to hypertension, unstable angina, myocardial infarction within the last 4 months, and uncontrolled congestive heart failure
* Cohort 2: Co-morbid illnesses or other concurrent disease, which in the judgment of the clinician obtaining informed consent, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Cohort 2: Patients with an ANC < 1.7 within 30 days of consent
* Cohort 2: Patients with an INR > 1.3 within 30 days of consent
* Cohort 2: Patients with a platelet count < 50 K, within 30 days of consent
* Cohort 2: Patients currently being treated with chemotherapy or within the preceding 30 days at the time of consent
* Cohort 2: Patients previously treated with a sacral nerve stimulator for urinary or fecal incontinence
* Cohort 2: Patients with an ECOG performance status > 2 at the time of consent
* Cohort 2: Patients with an active infection requiring systemic therapy at the time of consent
* Cohort 2: Patients with a significant history of uncontrolled cardiac disease including, but not limited to hypertension, unstable angina, myocardial infarction within the last 4 months, and uncontrolled congestive heart failure
* Cohort 2: Patients with an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig A Messick, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Sacral Nerve Stimulation (SNS): Patients undergo scheduled, elective surgery for placement of the sacral nerve stimulator with external battery pack. After 2 weeks, patients undergo implantation of a subcutaneous internal battery or removal of the leads if the sacral nerve stimulator is working but does not improve symptoms. If the sacral nerve stimulator is not working, it is repositioned and patients return 2 weeks later for implantation of external battery or removal of leads.
Period: Overall Study
Arm/Group | Experimental: Sacral Nerve Stimulation (SNS)
Started | 3
Completed | 1
Not Completed | 2
Not completed — Lack of Efficacy | 1
Not completed — Screen Failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: Sacral Nerve Stimulation (SNS)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Sacral Nerve Stimulation (SNS) Success
Description: SNS success will be measured as a patient having the battery implanted at visit 3. Patients who do not have the SNS placed, for any reason other than insurance coverage issues, will count as not having a success. Fecal incontinence will be measured by the physician as the total number of gas, mucus, liquid stool, and solid stool accidental leakage events reported in the bowel diaries. Improvement will be determined by the physician based on bowel diary comparisons recorded before SNS lead placement at visit 1 to after lead placement at visit 2. The proportion of patients who experience SNS success will be reported with a 90% credible interval using a beta (1,1)
Time Frame: Up to visit 3
Population: No data was collected
Arm/Group | Experimental: Sacral Nerve Stimulation (SNS)
Number analyzed (Participants) | 0

2. Secondary Outcome: Fecal Incontinence Severity Index Questionnaire Summary
Description: Will be reported descriptively with graphs or tabulations for categorical survey outcomes.
Time Frame: Up to 3 years
Population: No data was collected
Arm/Group | Experimental: Sacral Nerve Stimulation (SNS)
Number analyzed (Participants) | 0

3. Secondary Outcome: Fecal Incontinence Quality of Life Questionnaire Summary
Description: Will be reported descriptively with graphs or tabulations for categorical survey outcomes.
Time Frame: Up to 3 years
Population: No data was collected
Arm/Group | Experimental: Sacral Nerve Stimulation (SNS)
Number analyzed (Participants) | 0

4. Secondary Outcome: Euroqol-5 Dimensions-5 Levels (EQ-5D-5L)
Description: Will be reported descriptively with graphs or tabulations for categorical survey outcomes.
Time Frame: Up to 3 years
Population: No data was collected
Arm/Group | Experimental: Sacral Nerve Stimulation (SNS)
Number analyzed (Participants) | 0

5. Secondary Outcome: International Consultation on Incontinence Society - Female Lower Urinary Tract Symptoms
Description: Will be reported descriptively with graphs or tabulations for categorical survey outcomes.
Time Frame: Up to 3 years
Population: No data was collected
Arm/Group | Experimental: Sacral Nerve Stimulation (SNS)
Number analyzed (Participants) | 0

6. Secondary Outcome: Memorial Sloan Kettering Cancer Center Bowel Function Questionnaire (BFQ)
Description: Will be reported descriptively with graphs or tabulations for categorical survey outcomes.
Time Frame: Up to 3 years
Population: No data was collected
Arm/Group | Experimental: Sacral Nerve Stimulation (SNS)
Number analyzed (Participants) | 0

7. Secondary Outcome: Low Anterior Resection Syndrome Score BFQ
Description: Will be reported descriptively with graphs or tabulations for categorical survey outcomes.
Time Frame: Up to 3 years
Population: No data was collected
Arm/Group | Experimental: Sacral Nerve Stimulation (SNS)
Number analyzed (Participants) | 0

8. Secondary Outcome: Cleveland Clinic Incontinence Score
Description: Will be reported descriptively with graphs or tabulations for categorical survey outcomes.
Time Frame: Up to 3 years
Population: No data was collected
Arm/Group | Experimental: Sacral Nerve Stimulation (SNS)
Number analyzed (Participants) | 0

9. Secondary Outcome: Impact of SNS on Bowel Dysfunction
Description: Will be measured using bowel diaries.
Time Frame: Up to 30 days (visit 2)
Population: No data was collected
Arm/Group | Experimental: Sacral Nerve Stimulation (SNS)
Number analyzed (Participants) | 0

10. Secondary Outcome: Impact of SNS on Urinary Incontinence
Description: Will be measured using bladder diaries and a post-void urinary bladder residual and validated urinary symptom questionnaire.
Time Frame: Up to 30 days (visit 2)
Population: No data was collected
Arm/Group | Experimental: Sacral Nerve Stimulation (SNS)
Number analyzed (Participants) | 0

11. Secondary Outcome: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Colorectal 29
Description: Will be reported descriptively with graphs or tabulations for categorical survey outcomes.
Time Frame: Up to 3 years
Population: No data was collected
Arm/Group | Experimental: Sacral Nerve Stimulation (SNS)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From visit 1, up to 3 years
Arm/Group | Experimental: Sacral Nerve Stimulation (SNS)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/94/NCT04066894/Prot_SAP_000.pdf